CLINICAL TRIAL: NCT02701712
Title: Receiving Radiation Therapy in the MRgRT Research Facility
Acronym: MRgRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-8210-CE
Record Dates: First submitted 2016-02-22; First posted 2016-03-08 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumors and Metastatic Lesions
Keywords: magnetic resonance; external beam radiotherapy; brachytherapy; radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magnetic resonance - guided radiation therapy (MRgRT) (Experimental): Magnetic resonance (MR) - guided radiation therapy
  Interventions: Radiation: Magnetic resonance - guided radiation therapy (MRgRT)

INTERVENTIONS:
Radiation: Magnetic resonance - guided radiation therapy (MRgRT) — Use of magnetic resonance (MR) visualization for interventional radiotherapy in cancer patients

SUMMARY:
The aim of this study is to evaluate the technical performance of magnetic-resonance guided radiotherapy (MRgRT) facility at the Princess Margaret Cancer Centre and the impact on the workflow of the clinical team in this facility.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Planned to receive clinical intervention (imaging or treatment) in the MRgRT facility
* At least 18 years of age

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of planned patients receiving treatment in the MRgRT facility | 2 years

SECONDARY OUTCOMES:
Measure tumor size before, during and after radiotherapy | 2 years
  Collect and analyze imaging data before, during and after radiotherapy, and the related treatment data

CONTACTS AND LOCATIONS:
Overall Officials: Michael Milosevic, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada